CLINICAL TRIAL: NCT03002415
Title: Randomized Clinical Trial to Evaluate the Effect of Water Intake on the State of Hydration and Renal Function in Elderly Patients
Brief Title: The Effect of Water Intake on the State of Hydration and Renal Function in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 160153
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Renal Function Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided water intake (Experimental): Verbal and written guidelines will be given for the patient to ingest the daily volume of water calculated by the weight (30 ml / kg / day) for 14 days. Patients will receive an acrylic glass with a mark in 200 ml and will be instructed to take the number of glasses a day corresponding to the calculated volume (30 ml / kg). Patients will also receive a leaflet indicating how many glasses of water they will need to take. They will also be instructed to mark with an "X" the number of glasses of water that they actually drank daily during the fourteen days of intervention.
  Patients are asked to note on a food record food and liquids and quantities consumed throughout the day. Patients are advised to make a four-day food diary out of the 14 days.
  Interventions: Other: Guided water intake
- Placebo - free demand water intake (Placebo Comparator): Patients are instructed to drink water and other liquids on demand. Patients are asked to note on a food record food and liquids and quantities consumed throughout the day. Patients are advised to make a four-day food diary out of the 14 days.
  Interventions: Other: Placebo - free demand water intake

INTERVENTIONS:
Other: Guided water intake — Verbal and written guidelines will be given for the patient to ingest the daily volume of water calculated by the weight (30 ml / kg / day) for 14 days. Patients will receive an acrylic glass with a mark in 200 ml and will be instructed to take the number of glasses a day corresponding to the calculated volume (30 ml / kg). Patients will also receive a leaflet indicating how many glasses of water they will need to take. They will also be instructed to mark with an "X" the number of glasses of water that they actually drank daily during the fourteen days of intervention.
  Arms: Guided water intake
Other: Placebo - free demand water intake — Patients are instructed to drink water and other liquids on demand. Patients are asked to note on a food record food and liquids and quantities consumed throughout the day. Patients are advised to make a four-day food diary out of the 14 days.
  Arms: Placebo - free demand water intake

SUMMARY:
Acute dehydration in the elderly is a well-known clinical condition, although situations that lead to chronic dehydration in the elderly may be quite frequent, but they are poorly studied. Metabolic changes in body water homeostasis can influence and provide chronic dehydration status as reduced sensitivity to thirst, antidiuretic hormone and renal inability to concentrate urine and the presence of chronic diseases and the use of polypharmacy may also predispose states of chronic dehydration. Due to these facts, a study to detect the existence of chronic dehydration states in a population of elderly people is highly justifiable. In addition, understanding whether increased water intake, improving chronic dehydration, may improve renal function in this population seems to be of great value, since it is a simple and inexpensive intervention and, if confirmed, it can be taken to institutions, by family members and health promoters who care for and cohabit with elderly individuals.

Our main objective is to evaluate the effect of stimulated and calculated water intake (per kg of patient weight) on the state of hydration and renal function in a population of elderly individuals. It is also within the scope of this project to evaluate the presence of chronic dehydration in elderly patients as well as in a subgroup of diabetic patients, and to compare different methods of evaluation of renal function. Design: Clinical trial Randomized for the main objective and cross-sectional study for secondary objectives.

The principal hypothesis is that guided water intake improve renal function in elderly patients.

DETAILED DESCRIPTION:
Intervention:

Verbal and written guidelines will be given for the patient to ingest the daily volume of water calculated by the weight (30 ml / kg / day) for 14 days. Patients will receive an acrylic glass with a mark in 200 ml and will be instructed to take the number of glasses a day corresponding to the calculated volume (30 ml / kg). Patients will also receive a leaflet indicating how many glasses of water they will need to take. They will also be instructed to mark with an "X" the number of glasses of water that they actually drank daily during the fourteen days of intervention.

Measurements tools (applied on the first and second visits)

* Laboratory tests: serum and urinary osmolality, sodium, urea and serum creatinine. To evaluate the effect of hydration on the glycemic control of diabetic patients, the measurement of fasting glycaemia and glycated hemoglobin (enzymatic method and HCLP) will also be performed. These dosages will be performed at the HCPA Clinical Pathology Laboratory.
* Non-invasive test: electrical bioimpedance (BIA) InBody 370® will be used to evaluate the amount of free water, since it is simple, low cost and easy to perform in the outpatient clinics of elderly patients.
* Nutritional assessment: the MAN questionnaire (Mini nutritional assessment) will be applied to patients selected for the study at the first and second visits. Since a valid questionnaire to evaluate only water intake was not found, the MAN questionnaire was chosen because it contains questions related to water intake and because it is easy and quick to apply.
* MiniMental: The MiniMental cognitive function test will be applied on the first visit and after the observation period (second visit). The questionnaire is valid for the screening of cognitive disorders and it is a simple and quick method to evaluate the mental abilities of the patients under study.
* Food record: these are sheets with space designated for filling with food and liquids and quantities consumed throughout the day. Patients are advised to make a four-day food diary out of the 14 days.

Renal function will be assessed by estimation formulas (as recommended by NKF and KDIGO) that use serum creatinine (CKD-EPI, MDRD and BIS2) and formulas that use cystatin C (CKD- EPI-cys and BIS 1).

The assessment of GFR by 51Cr-EDTA will be performed in a subgroup of 15 patients from each arm of the study in a parallel manner before and after the intervention using the 51Cr-EDTA intravenous single injection technique at a dose of 150μCi with blood samples taken at 2, 3 and 4 hours later. Samples will be centrifuged and 2 ml of plasma will be pipetted in duplicate for gamma counter counting. An exponential equation evaluates the plasma decay of 51 Cr-EDTA, providing the value of GFR .

Serum creatinine will be determined by the calibrated Jaffe method (Roche), traceable to isotopic dilution mass spectrometry (ID-MS), with kinetic reading to minimize interference by bilirubin. The dosage of cystatin C will be performed by the immunoturbidimetry method (Roche). The coefficients of intra and interassay variation are 2.2% and 5.3%, respectively.

ELIGIBILITY:
Inclusion Criteria: Patients are eligible if they are 65 years-old or older, attend the department of Internal Medicine and Geriatrics of Hospital de Clínicas de Porto Alegre as outpatient and accept to participate in the study.

Exclusion Criteria: Patients will be excluded if they have heart failure NYHA class III and IV, pectoris angina and/or acute myocardial infarction in the last 3 months, pacemaker or implantable cardioverter defibrillator, stage 4 or 5 chronic renal failure (GFR <30ml / min / 1.73 m²), organic or cognitive impairment that unable the patients to ingest liquids, cirrhosis, and not compensated thyroid dysfunction.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Renal function Improvement by CKD-EPI formula | 14 days
  Renal function will be assess before and after 14 days of guided water intake on the intervention group and control group. CKD-EPI is a formula that considers serum creatinine, age, gender and race to estimate glomerular filtration rate.
Renal function Improvement by MDRD formula | 14 days
  Renal function will be assess before and after 14 days of guided water intake on the intervention group and control group. MDRD is a formula that considers serum creatinine, age, gender and race to estimate glomerular filtration rate.
Renal function Improvement by BIS-2 formula | 14 days
  Renal function will be assess before and after 14 days of guided water intake on the intervention group and control group. BIS-2 is a formula that considers serum creatinine and cystatin-C to estimate glomerular filtration rate.

SECONDARY OUTCOMES:
Assess dehydration measuring the free corporal water | 14 days
  Non-invasive test: electrical bioimpedance (BIA) InBody 370® will be used to evaluate the amount of free water, since it is simple, low cost and easy to perform in the outpatient clinics of elderly patients.
Assess if guided water intake can improve cognition | 14 days
  MiniMental: The MiniMental cognitive function test will be applied on the first visit and after the observation period. The questionnaire is valid for the screening of cognitive disorders and it is a simple and quick method to evaluate the mental abilities of the patients under study.
Assess the average amount of liquids taken by patients | 4 days
  Food record: sheets with space designated for filling with food and liquids and quantities consumed throughout the day. Patients are advised to make a four-day food diary out of the 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bauer, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided